CLINICAL TRIAL: NCT02780999
Title: Effect of Immobilization of the Metacarpophalangeal Joint in Thumb Osteoarthritis on Pain and Function Three Months Follow up: Randomized Clinical Trial
Brief Title: Effect of Immobilization of the Metacarpophalangeal Joint in Thumb Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Raquel Cantero-Téllez, Profesor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19761
Record Dates: First submitted 2016-05-10; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Hand Osteoarthritis
Keywords: Osteoarthritis; hand; orthotic; rehabilitation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): It is a thumb orthotic that does not include wrist joint but includes the metacarpophalangeal joint.
  Interventions: Device: Whale orthosis
- Control group (Active Comparator): It is a thumb orthotic that does not include wrist joint neither metacarpophalangeal joint.
  Interventions: Device: Colditz orthosis

INTERVENTIONS:
Device: Whale orthosis — Participants will be teach how to use the Whale orthotic to be carried for a period of three months during night and during the day in dose activities that cause pain
  Arms: Experimental group
Device: Colditz orthosis — Participants will be teach how to use the Colditz orthotic to be carried for a period of three months during night and during the day in dose activities that cause pain.
  Arms: Control group

SUMMARY:
The aim of this study is to compare the effect of Whale and Colditz static orthosis on pain and functional abilities of hand in thumb carpometacarpal osteoarthritis as a unique treatment.

Patients with thumb CMC OA will be recruited at Tecan Hand Center Clinic. Participants will be assigned using a randomized allocation in two groups. For group A a "Whale orthotic" will be constructed and for group B a Colditz orthotic. Both static splint will endorse for 3 months. Inclusion criteria for this study were adult over 18 diagnosed with carpometacarpal joint osteoarthritis with a pain intensity during Activities of Daily Living (ADL's) up to 4 / 10 on the Visual Analog Scale (VAS).

Patients were excluded from participation if they had: a neurological disorder affecting the upper limb; had received previous treatment for their hand problem in the last 6 months including an intra-articular joint injection to wrist, fingers or thumb; had fractures or a significant hand injury or previous surgery to the wrist or hand; had hand or finger tenosynovitis and/ or Dupuytren's disease. Were also excluded patients who did not complete Dash Spanish version questionnaire or if they did not sign the informed consent.

The outcome measure will be pain intensity and functional abilities as measured with the Visual Analogue Scale (VAS) and Disabilities of the Arm, Shoulder and Hand (DASH), respectively. All measures will be collected at baseline and end of the intervention.

DETAILED DESCRIPTION:
A hand therapy blinded to the subjects' intervention took baseline measurements (Spanish- Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire and pain intensity) prior to randomization.

Participants were introduced in an Excel database in order of arrival and were randomized into 2 equal groups by an automatic program (Group A : Whale orthotic. Group B Colditz Orthotic). The same low temperature thermoplastic material was used for both orthoses (Orfit Colors NS 2.0 mm, micro perforated/ Orfit Industries, Wijnegem, Belgium). The orthoses were custom -fabricated for each patient by a hand therapy clinician experienced in orthopedic cases.

Both groups of patients received identical orthotic wearing instructions. Patients were asked to use the orthosis during the nighttime and also during daytime ADL's for three to four hours per day. Each patient was also provided with a data collection sheet in order to control treatment adherence. All patients were asked to report any discomfort when using the orthosis. The orthosis was the only treatment intervention received by the participants. No therapeutic exercises, modalities or other complementary treatments were offered to the patients in order not to interfere with the individual effectiveness of the orthosis. Patients were contacted by telephone a week after and were ask about pain intensity. Three months after first evaluation, participants were cited in hand therapy clinic in order to collect again outcomes measurements.

ELIGIBILITY:
INCLUSION CRITERIA:

* 18 years old
* Having diagnosed with carpometacarpal joint osteoarthritis
* Had given their consent

EXCLUSION CRITERIA:

* Had neurological disorder affecting the upper limb
* Had received previous treatment for their hand problem in the last 6 months
* Had hand or finger tenosynovitis
* Suffering Dupuytren's disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of Pain intensity | Change from Baseline and at 3-month post-interventions
  Visual analogue scale

SECONDARY OUTCOMES:
Change of DASH questionnaire | Change from Baseline and at 3-month post-interventions
  Upper limb function

CONTACTS AND LOCATIONS:
Overall Officials: Cantero-Tellez Raquel, PhD, Principal Investigator — University of Malaga
Locations (1):
- Raquel Cantero-Téllez, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cantero-Tellez R, Villafane JH, Valdes K, Berjano P. Effect of immobilization of metacarpophalangeal joint in thumb carpometacarpal osteoarthritis on pain and function. A quasi-experimental trial. J Hand Ther. 2018 Jan-Mar;31(1):68-73. doi: 10.1016/j.jht.2016.11.005. Epub 2017 Feb 22. PMID 28237072